CLINICAL TRIAL: NCT00558675
Title: A Phase I/II Study of Intentionally Mis-Matched, Allogeneic Th1 Memory Cells (AlloStim) Conjugated With CD3/CD28-coated Microbeads in Patients With Relapsed or Refractory Hematological Malignancy
Brief Title: A Phase I/II Study of Mis-Matched Immune Cells (AlloStim) in Patients With Advanced Hematological Malignancy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mirror Biologics, Inc. (Industry)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITL-001-HMC
Record Dates: First submitted 2007-11-13; First posted 2007-11-15 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2012-11

CONDITIONS: Hematological Malignancy; Leukemia; Lymphoma; Multiple Myeloma
Keywords: Non-Hodgkins Lymphoma; Hodgkins Lymphoma; Acute Lymphoblastic Leukemia; Chronic Myeloid Leukemia; Chronic Lymphocytic Leukemia; Multiple Myeloma; Immunotherapy; Allogeneic Cell Therapy
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma; Multiple Myeloma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Single intravenous infusion of AlloStim
  Interventions: Biological: AlloStim
- 2 (Experimental): Intravenous AlloStim infusion on day 1 and day 7
  Interventions: Biological: AlloStim
- 3 (Experimental): Intravenous AlloStim infusion on day 1, day 7 and day 14
  Interventions: Biological: AlloStim
- 4 (Experimental): Intravenous AlloStim infusion on day 1, day 7, day 14 and day 21
  Interventions: Biological: AlloStim

INTERVENTIONS:
Biological: AlloStim — single intravenous infusion of 1 x 10^9 AlloStim cells
  Arms: 1
Biological: AlloStim — Intravenous infusion of 1 x 10^9 AlloStim on day 1 and a second intravenous infusion of 1 x 10^8 AlloStim on day 7
  Arms: 2
Biological: AlloStim — Intravenous infusion of 1 x 10^9 AlloStim on day 1 and a second intravenous infusion of 1 x 10^8 AlloStim on day 7 and day 14
  Arms: 3
Biological: AlloStim — Intravenous infusion of 1 x 10^9 AlloStim on day 1 and a second intravenous infusion of 1 x 10^8 AlloStim on day 7, day 14 and day 21
  Arms: 4

SUMMARY:
The purpose of this study is to determine the safety and anti-tumor effects of an experimental immunotherapy drug, called AlloStim, which is intentionally mis-matched immune cells which are designed to elicit the same anti-tumor mechanism that occurs in allogeneic bone marrow/stem cell mini-transplant (BMT) procedures, without the toxicity associated with graft vs. host disease (GVHD).

DETAILED DESCRIPTION:
AlloStim is combination biological drug and medical device formulation consisting of allogeneic immune cells that have been expanded and differentiated ex-vivo. These cells are conjugated to monoclonal antibody coated microparticles prior to infusion. The immune cells are living CD4+ memory Th1-like T-cells (T-Stim) that are differentiated from precursors purified from normal donor blood. AlloStim is a composition of T-Stim cells conjugated to paramagnetic epoxy covered microparticles (4.5micron) with covalently bound anti-CD3/anti-CD28 monoclonal antibodies (Dynabeads® ClinExVivo™ CD3/CD28) at a 2:1 bead:cell ratio. The T-Stim cells are intentionally mismatched to the recipient.

The graft vs. tumor (GVT) effect that occurs after allogeneic bone marrow transplant (BMT) is a curative therapy for advanced hematological malignancy but the clinical application of GVT is severely limited by graft vs. host disease (GVHD) toxicity. AlloStim is designed to elicit the "mirror" of the GVT/GVHD effects in the host immune system. Rather than trying to separate these effects, we have proposed that the effects could remain associated and "mirrored" onto the host immune system creating linked host vs. tumor (HVT) and host vs. graft (HVG) effects. We hypothesized that allogeneic Th1 memory cells activated at time of infusion to produce type 1 cytokines and express CD40L would elicit HVT/HVG "mirror effects" in immunocompetent cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed hematological malignancy
* unresponsive to chemotherapy and/or recurrence after autologous transplant
* adequate kidney, liver, lung and heart function

Exclusion Criteria:

* prior allogeneic transplant
* immunosuppressive therapy for concurrent medical condition
* active viral infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Determination of toxicity related to AlloStim infusion in accordance with NCI Common Toxicity Criteria v.3 | Within first 48 hours post infusion, at 30 days and at 60 days post infusion

SECONDARY OUTCOMES:
Evaluation and reporting of anti-tumor response will be conducted in accordance with internationally accepted criteria for the disease indication being evaluated | 30 days and 60 days post infusion and yearly thereafter
Immunological Response | 30 days, 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Michael Har-Noy, Principal Investigator — Immunovative Therapies
Locations (1):
- Hadassah-Hebrew University Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Har-Noy M, Slavin S. The anti-tumor effect of allogeneic bone marrow/stem cell transplant without graft vs. host disease toxicity and without a matched donor requirement? Med Hypotheses. 2008;70(6):1186-92. doi: 10.1016/j.mehy.2007.10.008. Epub 2007 Dec 3. PMID 18054441
- [Background] Har-Noy M, Zeira M, Weiss L, Slavin S. Completely mismatched allogeneic CD3/CD28 cross-linked Th1 memory cells elicit anti-leukemia effects in unconditioned hosts without GVHD toxicity. Leuk Res. 2008 Dec;32(12):1903-13. doi: 10.1016/j.leukres.2008.05.007. Epub 2008 Jun 18. PMID 18565579
- [Background] Har-Noy M, Zeira M, Weiss L, Fingerut E, Or R, Slavin S. Allogeneic CD3/CD28 cross-linked Th1 memory cells provide potent adjuvant effects for active immunotherapy of leukemia/lymphoma. Leuk Res. 2009 Apr;33(4):525-38. doi: 10.1016/j.leukres.2008.08.017. Epub 2008 Oct 1. PMID 18834631